CLINICAL TRIAL: NCT05769075
Title: A Phase I, Multicenter, Open-label Study of TY-2136b, Administered Orally in Patients With Advanced or Metastatic Solid Tumors Harboring ALK, ROS1 or NTRK1-3 Alterations
Brief Title: A Study of TY-2136b in Patients With Advanced Solid Tumors Harboring ALK, ROS1 or NTRK1-3 Alterations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TYKM7203101
Record Dates: First submitted 2023-02-09; First posted 2023-03-15 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escalation stage (Experimental): Escalation stage: Multiple doses of TY-2136b for oral administration to find the maximum tolerated dose
  Interventions: Drug: TY-2136b
- Expansion stage (Experimental): Expansion stage: 4 distinct expansion cohorts
  Interventions: Drug: TY-2136b

INTERVENTIONS:
Drug: TY-2136b — Drug: TY-2136b PO, QD or BID
  Escalation stage: 7 increased dose cohorts from low dose to MTD (from 40mg QD to 420mg QD)
  Arms: Escalation stage
Drug: TY-2136b — Expansion stage: 4 distinct cohorts
  The dose for the Expansion stage will be determined based on results from the Escalation stage
  Arms: Expansion stage

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of TY-2136b and to determine the recommended phase 2 dose (RP2D), with dose-escalation stage and dose-expansion stage.

DETAILED DESCRIPTION:
* To evaluate the pharmacokinetic (PK) characteristics of TY-2136b after single and multiple oral doses.
* To assess preliminary antitumor activity of TY-2136b as a single agent when administered orally to patients with advanced or metastatic solid tumors.
* To identify mutations in the ALK, ROS1 and NTRK1-3, or other molecular alterations in blood or tumor tissues associated with clinical outcome.

ELIGIBILITY:
Inclusion criteria:

1. Willing and able to provide written informed consent approved by institutional review board (IRB) or independent ethics committee (IEC).
2. In the escalation stage, patients should fulfill the following criterion at Screening:

   1. Age ≥18 years.
   2. Histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumor. Evidence of ALK, ROS1, NTRK1, NTRK2 or NTRK3 alterations in tumor tissue or blood, as determined with prior molecular assays performed in a CLIA-certified or equivalent laboratory.
   3. Patients must have failed established standard medical anti-cancer therapies for a given tumor type or have been intolerant to such therapy, or in the opinion of the Investigator have been considered ineligible for a particular form of standard therapy on medical grounds. Note: Prior cytotoxic chemotherapy is allowed; prior anti-cancer immunotherapy is allowed.

   In the expansion stage, patients should fulfill the following criteria at Screening:
   1. Age ≥18 years.
   2. Histologically or cytologically confirmed diagnosis of locally advanced or metastatic NSCLC and other solid tumors.
   3. Subject must have a documented ROS1 or NTRK1-3 gene or ALK fusion or rearrangement determined by CLIA-certified or equivalent testings. Next-generation sequencing (NGS), quantitative polymerase chain reaction (qPCR) test or fluorescence in situ hybridization (FISH).
3. ECOG Performance Status 0-1.
4. Capability to swallow intact tablet without chewing or opening; if the patient cannot swallow many tablets of high dose at one time, the subject can take dissolving tablets orally.
5. At least 1 measurable target lesion according to Response Evaluation Criteria in Solid Tumor Version 1.1 (RECIST v1.1) determined by the investigator. Subjects with central nervous system (CNS)-only measurable disease ≥10 mm as defined by RECIST v1.1 are eligible.
6. All acute toxic effects (excluding alopecia of any prior anticancer therapy recovered to grade ≤1 based on NCI CTCAE v5.0).
7. Patients with asymptomatic CNS metastases (treated or untreated) are also eligible if they satisfy the other criteria specified in this protocol.
8. Baseline laboratory results fulfilling the requirements.
9. Life expectancy ≥3 months.
10. For female patients of childbearing potential, the serum or urine pregnancy test within 72 hours prior to the start of TY-2136b treatment should be negative.
11. Male and female patients of childbearing potential must agree to use 2 methods of highly effective contraception from signing ICF, throughout the study and continued for 90 days after the last dose of TY-2136b treatment.
12. Willing and able to comply with all aspects of the protocol.

Exclusion criteria:

1. Concurrent participation in another therapeutic clinical trial. Unless the patient is during follow-up period of a previous interventional clinical trial.
2. Symptomatic CNS metastases, OR leptomeningeal involvement.
3. History of other previous cancer (except for squamous cell or basal-cell carcinoma of the skin, any in situ carcinoma that has been completely resected, or other early-stage malignancies receiving curative treatment which get consensus between the investigators and sponsor), requiring therapy within the previous 2 years.
4. Major surgery within 4 weeks prior to the start of TY-2136b treatment; OR radiation therapy (except palliative to relieve bone pain) within 2 weeks prior to enrollment. Note: Palliative radiation must have been completed at least 48 hours prior to enrollment.
5. Patients receiving long-term systemic immunosuppressant therapy (≤10 mg/ day of prednisone or another equivalent dose of corticosteroid inhalation or topical administration can be included);
6. Clinically significant cardiovascular disease (either active at Screening or within 6 months prior to enrollment): myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association Classification Class ≥II), cerebrovascular accident or transient ischemic attack, stroke, symptomatic bradycardia, or requirement for anti-arrhythmic medication; or cardiac dysrhythmias of NCI CTCAE grade ≥2 deemed of clinical significance by the investigator.
7. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (electrocardiogram interval measured from the onset of the QRS complex to the end of the T wave) for heart rate (QTcF) >470 msec obtained from 3 electrocardiograms, using the screening clinic electrocardiogram machine derived QTc value.
   2. Any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiogram (e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec).
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or any concomitant medication known to prolong the QT interval during Screening.
8. Known active infections, e.g., bacterial, fungal and viral infections, including human immunodeficiency virus (HIV) infection (defined as anti-HIV antibody positive), hepatitis B virus (HBV) infection [defined as Hepatitis B surface antigen (HBsAg) positive and HBV-DNA ≥1000 cps/mL or 200 IU/mL] and hepatitis C virus (HCV) infection (defined as anti-HCV antibody positive and HCV-RNA positive). Human Immunodeficiency Virus (HIV) positive patients could be eligible after discussion with medical monitor based on current and past CD4 and T-cell counts, history (if any) of AIDS-defining conditions (e.g., opportunistic infections), and status of HIV treatment.
9. Active gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, short gut syndrome) or other malabsorption syndromes that will impact drug absorption.
10. Peripheral neuropathy of CTCAE ≥ grade 2.
11. History of extensive, disseminated, bilateral or CTCAE grade 3 or 4 interstitial fibrosis or interstitial lung disease (ILD) including pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, ILD, obliterative bronchiolitis, and pulmonary fibrosis. Note: Patients with history of prior radiation pneumonitis will not be excluded.
12. History of strong inhibitors and/or inducers of CYP3A within 2 weeks prior to the first dose of TY-2136b.
13. History of strong inhibitors and/or inducers of P-glycoprotein within 2 weeks prior to the first dose of TY-2136b.
14. History of sensitive substrates and those with a narrow therapeutic index of CYP2C8, CYP2C9, CYP2C19, CYP2D6 and CYP3A within 2 weeks prior to the first dose of TY-2136b.
15. History of proton pump inhibitors (PPIs) within 4 days prior to the first dose of TY-2136b; OR history of histamine H2 blockers within 2 days prior to the first dose of TY-2136b.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
(Escalation stage) Dose Limiting Toxicities (DLTs) | Within 28 days of the first dose
  Numbers of participants experiencing AEs which are defined as DLTs classfied by CTCAE v5.0.
(Escalation stage) Recommended Phase 2 Dose (RP2D) | Within 28 days of the last patient dosed in escalation stage
  The RP2D is defined as the dose level chosen for the dose expansion arms, based on safety, tolerability, efficacy, pharmacokinetics (PK), and pharmacodynamic (PD) data collected during the dose escalation portion of the study.
(Escalation stage) Adverse events (AEs) | From Baseline up to 28 days after the end of the treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
(Expansion stage) Overall Response Rate (ORR) | From the date of first dose until the date of first documented progression or stable disease or the date of death from any cause, whichever came first, assessed up to 30 months.
  ORR is defined as the percentage of subjects who have a partial response (PR) or complete response (CR) to the treatment response assessment in accordance to Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

SECONDARY OUTCOMES:
(Escalation and Expansion stage) Area under the plasma concentration time curve(AUC0-inf) | Cycle 1 Day 1 (at pre-dose, 0.5, 1, 2, 4, 6, 24 h post-dose) (Each Cycle=28 days)
  AUC0-inf defined as the area under the plasma concentration-time curve from time 0 extrapolated to Infinite time.
(Escalation and Expansion stage) Area under the plasma concentration time curve(AUC0-t) | Cycle 1 Day 1 and Cycle 1 Day 21 (at pre-dose, 0.5,1, 2, 4, 6, 24 hours post-dose)(Each Cycle=28 days)
  AUC0-t defined as area under the plasma concentration-time curve from time 0 to time t.
(Escalation and Expansion stage) Maximum plasma concentration (Cmax) | Cycle 1 Day1 and Cycle 1 Day 21 (at pre-dose, 0.5,1, 2, 4, 6, 24 hours post-dose)(Each Cycle=28 days)
  Cmax is the maximum (or peak) plasma concentration that the drug achieves in blood after the drug has been administered.
(Escalation and Expansion stage) Minimum plasma concentration (Cmin) | Cycle1 Day 21 (at pre-dose, 0.5,1, 2, 4, 6, 24 hours post-dose)(Each Cycle=28 days)
  Cmin is the minimum plasma concentration that the drug achieves in blood after the drug has been administered.
(Escalation and Expansion stage) Terminal half-life (t1/2) | Cycle1 Day 1 and Cycle1 Day 21 (at pre-dose, 0.5,1, 2, 4, 6, 24 hours post-dose)(Each Cycle=28 days)
  T1/2 is defined as the time for the concentration of a compound in sytemic circulation to reduce by half.
(Escalation and Expansion stage) The time to the peak concentration (Tmax) | Cycle1 Day 1 and Cycle1 Day 21 (at pre-dose, 0.5,1, 2, 4, 6, 24 hours post-dose)(Each Cycle=28 days)
  Tmax is defined as the time of maximum concentration of the drug in blood observed after a drug dose administration.
(Escalation and Expansion stage) Progression-free survival (PFS) | Up to 30 months after the date of first dose.
  PFS is defined as the time from randomization until first evidence of disease progression or death.
(Escalation and Expansion stage) Duration of Response (DOR) | Up to 30 months after the date of first dose.
  DOR is defined as the time from randomization to disease progression or death in patients who achieve complete or partial response.
(Escalation and Expansion stage) Overall survival (OS) | Up to 30 months after the date of first dose.
  OS is defined as the time from the start of treatment to death or the end of the study.
(Escalation stage) Overall Response Rate (ORR) | From the date of first dose until the date of first documented progression or stable disease or the date of death from any cause, whichever came first, assessed up to 30 months.
  ORR is defined as the percentage of subjects who have a partial response (PR) or complete response (CR) to the treatment response assessment in accordance to Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: TYK Medicines, Inc, Study Director — TYK Medicines, Inc
Locations (2):
- United States (2):
  - Rhode Island Hospital, Brown University, Providence, Rhode Island
  - Oncology Consultants, Houston, Texas

IPD SHARING:
Plan to Share IPD: No